CLINICAL TRIAL: NCT03805750
Title: A Double-Blind, Cross-Over, Placebo- Controlled Efficacy and Tolerability Study of Oral Cannabidiol (CBD) and Tetrahydrocannabinol (THC) for Essential Tremor (ET).
Brief Title: Trial of Cannabis for Essential Tremor
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: International Essential Tremor Foundation (Other); Tilray (Industry); Center for Medicinal Cannabis Research (Other)
Responsible Party: Principal Investigator, Fatta B Nahab, Associate Professor of Neurosciences, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 180414
Record Dates: First submitted 2019-01-09; First posted 2019-01-16 (Actual); Results first posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor | interventions — nabiximols; Cannabidiol; Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CBD/THC (Experimental): Treatment arm consisting of Tetrahydrocannabinol (5mg/capsule) and Cannabidiol (100mg/capsule).
  Interventions: Drug: CBD/THC
- Placebo (Placebo Comparator): Matched placebo capsule with no active ingredients.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: CBD/THC — Oral formulation of combined Cannabidiol (CBD) and Tetrahydrocannabinol (THC).
  Other Names: marijuana; cannabis; cannabidiol; tetrahydrocannabinol
  Arms: CBD/THC
Drug: Placebo oral capsule — Matched Placebo
  Arms: Placebo

SUMMARY:
This is a pilot trial to evaluate the safety and efficacy of a combined oral formulation of THC and CBD in patients with Essential Tremor.

DETAILED DESCRIPTION:
Essential tremor (ET) is the most common neurological movement disorder, affecting up to 1% of the population and up to 5% of individuals over the age of 65. ET is characterized by often disabling tremors that occur when an individual moves. The tremors most commonly affect the hands, head, voice, and legs in order of frequency, leading to impairment in activities of daily living and morbidity. No pharmacological agent has been developed for ET, though existing agents such as propranolol and primidone are used off-label to reduce tremor amplitude. Deep brain stimulation surgery is often reserved for only individuals with the most severe tremors. Patients with ET have long reported tremor benefits with the use of cannabis, though no controlled trials have been conducted. The investigators plan to conduct the first double-blind, placebo-control clinical trial of cannabis in an oral capsule. Various validated tremor rating methods will be used to quantify tremor severity, while looking at tolerability and safety.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ET by a Movement Disorder Neurologist
* Stable dose of tremor medication for a period of at least 6 weeks prior to screening
* Tremor in the arms
* Tremor(s) is/are moderately severe (amplitude of at least 1cm)

Exclusion Criteria:

* Significant non-ET related abnormal findings on neurological exam
* Tremor at rest, or other features suggestive of Parkinson disease
* Diagnosis of dementia
* Pregnant or nursing
* Childbearing potential and unable or unwilling to use contraception during course of the trial
* On medications known to interact with the study drug
* Current or prior history of alcohol or substance abuse
* Recent exposure to primidone (within the past 21 days) or benzodiazepines (such as Valium, Ativan or Klonopin), ketoconazole, ritonavir, clarithromycin, rifampin, carbamazepine, St. Johns Wort, digoxin or other medications known to affect your liver enzymes (within the past 7 days).
* Unwilling to abstain from consuming grapefruits, grapefruit juice or grapefruit containing products.
* Taking medications such as warfarin, cyclosporine, and amphotericin B that are highly protein-bound
* Do not wish to take a cannabis-derived agent
* Allergy or sensitivity to sorbitol, xylitol, stevia or other natural sweeteners
* Allergy or sensitivity to cannabis
* Used cannabis or a cannabis-derived product (such as CBD oil) within the past 4 weeks or plan to use it during this research study.
* Diagnosis of a psychiatric disorder (e.g., mania, bipolar depressive disorder, schizophrenia, schizoaffective disorder, or other major psychiatric disorder)
* Current or prior history of suicidal thoughts and/or behavior
* Active medical problem affecting the immune system, liver, gastrointestinal tract, lungs, heart, endocrine system (such as diabetes and/or thyroid), and/or a blood clotting disorder
* Current infection
* Reduced kidney function (GFR <60)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fatta Nahab, MD, Principal Investigator — UCSD
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Information — http://tremor.cmcr.ucsd.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a cross-over design where each subject receives both a placebo and treatment arm in blinded random order.
Groups:
- CBD/THC First Then Placebo; Placebo First Then CBD/THC: After randomization, each patient will receive study medication in two study periods. Each study period includes 1-week titration, 2-week treatment, and 1-week tapering. There is a 3-week washout period between the two study periods. During the titration period, patients will have a starting dose of 1 capsule (placebo or 5mg THC/100mg CBD) per day; 2 capsules per day on day 3; 3 capsules per day on day 6. If the patient or investigator feel that the higher study drug dose of 3 caps per day is causing troublesome side effects, the dosage may be lowered to 2 caps per day. Patients will continue on this target dose during the 2-week treatment and then gradually taper from medication over one week. Patients will crossover to the alternate treatment after a 3-week washout period.
Period: First Intervention - 4 Weeks
Arm/Group | CBD/THC First Then Placebo | Placebo First Then CBD/THC
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0
Period: Second Intervention - 4 Weeks
Arm/Group | CBD/THC First Then Placebo | Placebo First Then CBD/THC
Started | 3 | 4
Completed | 3 | 2
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Participants: After randomization, each patient will receive study medication in two study periods. Each study period includes 1-week titration, 2-week treatment, and 1-week tapering. There is a 3-week washout period between the two study periods. During the titration period, patients will have a starting dose of 1 capsule (placebo or 5mg THC/100mg CBD) per day; 2 capsules per day on day 3; 3 capsules per day on day 6. If the patient or investigator feel that the higher study drug dose of 3 caps per day is causing troublesome side effects, the dosage may be lowered to 2 caps per day. Patients will continue on this target dose during the 2-week treatment and then gradually taper from medication over one week. Patients will crossover to the alternate treatment after a 3-week washout period.
Arm/Group | All Participants
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Digital Spirography
Description: The tremor mean amplitude calculated using computerized spirography to measure kinetic tremors.
Time Frame: Day 22 (100 minutes post-dose)
Measure: Mean (Standard Deviation); unit: millimeters of tremor amplitude
Groups:
- CBD/THC: Treatment arm
  CBD/THC: Oral formulation of CBD and THC.
- Placebo: Placebo oral capsule: Placebo
Arm/Group | CBD/THC | Placebo
Number analyzed (Participants) | 5 | 7
millimeters of tremor amplitude | 1.04 (0.57) | 1.00 (0.42)

2. Secondary Outcome: Change in Score on a Scale From Baseline of the Tremor Research Group Essential Tremor Rating Scale (TETRAS)
Description: The performance sub scale of the TETRAS will be used to measure tremor severity. The scale ranges from 0 to 60 points (0 being no tremor).
Time Frame: Baseline and Day 22
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBD/THC | Placebo
Number analyzed (Participants) | 5 | 7
score on a scale | -8.07 (5.71) | -10.3 (3.9)

3. Secondary Outcome: Global Impression of Change
Description: The Global impression of change will be calculated based on both physician and patient report. The scale ranges from a score of 1 (very much improved) to 7 (very much worse) with a score of 4 indicating 'no change'.
Time Frame: Day 22
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | CBD/THC | Placebo
Number analyzed (Participants) | 5 | 7
score on a scale
  Clinical Global Impression of Change | 3 [3 to 4] | 4 [2 to 4]
  Patient Global Impression of Change | 3 [3 to 4] | 4 [2.5 to 4]

4. Secondary Outcome: Number of Participants Reporting Adverse Events Based on Common Terminology Criteria
Description: Side effects survey
Time Frame: Days 1, 3, 6, 22
Measure: Count of Participants; unit: Participants
Arm/Group | CBD/THC | Placebo
Number analyzed (Participants) | 7 | 7
Participants
  Ringing in ears | 7 | 6
  Numbness/tingling | 4 | 4
  Dyspnea on exertion | 4 | 4
  Watery eyes | 3 | 3
  Runny nose | 3 | 2
  Decreased concentration | 7 | 0
  Sleepiness | 4 | 1
  Insomnia | 0 | 2
  Increased sleepiness | 2 | 1
  Dizziness | 4 | 0
  Memory problems | 3 | 0
  Imbalance | 3 | 0
  Mild headache | 0 | 1
  Groggy | 0 | 1
  Tired | 0 | 1
  Thumb pain | 0 | 1
  Anxiety | 2 | 0
  Headache | 2 | 0
  Lightheaded | 2 | 0
  Felt high | 1 | 0
  Decreased libido | 1 | 0
  Diarrhea | 1 | 0
  Dry mouth | 1 | 0
  Euphoria | 1 | 0
  Fatigue | 1 | 0
  Feels relaxed | 1 | 0
  Increased thirst | 1 | 0
  Felt buzzed | 1 | 0
  Quivering voice | 1 | 0
  Visual slowing | 1 | 0

5. Secondary Outcome: Number of Participants at Risk for Suicide Based on Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: This is a scale looking at risk assessment of suicidality. The presence of any positive responses will lead to further evaluation.
Time Frame: Day 22
Measure: Count of Participants; unit: Participants
Arm/Group | CBD/THC | Placebo
Number analyzed (Participants) | 5 | 7
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With New Study-related Electrocardiogram (EKG) Abnormalities
Description: Electrocardiographic changes from baseline measures will trigger further evaluation. EKG's will be rated as normal/abnormal relative to the baseline EKG reading, and abnormal findings will be rated as clinically significant/not clinically significant.
Time Frame: Day 22
Measure: Count of Participants; unit: Participants
Arm/Group | CBD/THC | Placebo
Number analyzed (Participants) | 5 | 7
Participants | 0 | 0
Statistical Analysis 1: Comparison: CBD/THC vs Placebo; Test type: Other; p = 0.52, Regression, Logistic

7. Secondary Outcome: Accelerometry-based Assessment of Tremor Severity
Description: The spectral power density measure of accelerometry data to measure will serve as a measure of tremor severity, comparing tremor amplitude from this digital biomarker at the time of the primary outcome to the same measure at baseline.
Time Frame: Baseline and Day 22
Population: Participants in both treatment arms will undergone tremor measurement using accelerometry as a surrogate of tremor severity.
Measure: Mean (Standard Deviation); unit: Proportion of baseline spectral power
Arm/Group | CBD/THC | Placebo
Number analyzed (Participants) | 5 | 7
Proportion of baseline spectral power | 0.012 (0.03) | 0.007 (0.011)

ADVERSE EVENTS:
Time Frame: Over the course of the study period (77 days).
Arm/Group | CBD/THC | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 7/7 | 6/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CBD/THC (N=7) | Placebo (N=7)
Ringing in ears (Ear and labyrinth disorders) | 7 | 6
Numbness/tingling (Nervous system disorders) | 4 | 4
Dyspnea on exertion (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Watery eyes (Eye disorders) | 3 | 3
Runny nose (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Decreased concentration (Nervous system disorders) | 7 | 0
Sleepiness (Nervous system disorders) | 4 | 1
Insomnia (Nervous system disorders) | 0 | 2
Increased sleepiness (Nervous system disorders) | 2 | 1
Dizziness (Nervous system disorders) | 4 | 0
Memory problems (Nervous system disorders) | 3 | 0
Imbalance (Nervous system disorders) | 3 | 0
Mild headache (Nervous system disorders) | 0 | 1
Grogginess/cognitive slowing (Nervous system disorders) | 0 | 1
Tiredness (Nervous system disorders) | 0 | 1
Thumb pain (Skin and subcutaneous tissue disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 0
Lightheadedness (Cardiac disorders) | 2 | 0
Feeling high/intoxication (Nervous system disorders) | 1 | 0
Decreased libido (General disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Euphoria (Psychiatric disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Feeling relaxed (General disorders) | 1 | 0
Increased thirst (Gastrointestinal disorders) | 1 | 0
Felt buzzed (Nervous system disorders) | 1 | 0
Quivering voice (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Visual slowing (Eye disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-09-30): https://cdn.clinicaltrials.gov/large-docs/50/NCT03805750/Prot_SAP_002.pdf